CLINICAL TRIAL: NCT03840278
Title: The Bihormonal iLet Bionic Pancreas Feasibility Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beta Bionics, Inc. (Industry); Zealand Pharma (Industry)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000252; 19-002 (Other: Zealand Pharma)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: bionic pancreas; closed loop; glucagon; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — dasiglucagon

STUDY DESIGN:
Intervention Model Description: The study follows a 2-treatment, 2-period crossover design, 2 and will consist of two 7-day study arms in random order: one bihormonal bionic pancreas arm using insulin lispro or insulin aspart and dasiglucagon, and one insulin-only bionic pancreas arm using insulin lispro or insulin aspart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Bihormonal iLet first, then Insulin-Only iLet (Experimental): Each sequence of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or dasiglucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM).
  For this sequence, participants first used the bihormonal iLet bionic pancreas for 1 week. They then used the insulin-only iLet bionic pancreas for 1 week.
  Interventions: Device: Bihormonal iLet Bionic Pancreas; Drug: Dasiglucagon
- Insulin-Only iLet first, then Bihormonal iLet (Experimental): Each sequence of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or dasiglucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM).
  For this sequence, participants first used the insulin-only iLet bionic pancreas for 1 week. They then used the bihormonal iLet bionic pancreas for 1 week.
  Interventions: Device: Insulin-only Bionic Pancreas

INTERVENTIONS:
Device: Bihormonal iLet Bionic Pancreas — Bihormonal iLet Bionic Pancreas using insulin and dasiglucagon
  Arms: Bihormonal iLet first, then Insulin-Only iLet
Device: Insulin-only Bionic Pancreas — Insulin-only iLet Bionic Pancreas using just insulin
  Arms: Insulin-Only iLet first, then Bihormonal iLet
Drug: Dasiglucagon — Experimental stable glucagon for use in the iLet Bionic Pancreas
  Arms: Bihormonal iLet first, then Insulin-Only iLet

SUMMARY:
Our objective is to evaluate the function of the bihormonal configuration of the ILet bionic pancreas delivering dasiglucagon when compared to the insulin-only configuration of the ILet bionic pancreas in a home-use study in adults with type 1 diabetes.

DETAILED DESCRIPTION:
Our objective is to conduct a home-use study testing the Gen 3.2 iLet bionic pancreas system in the insulin-only configuration and the bihormonal configuration with dasiglucagion in 10 adult subjects (≥ 18 years old) with type 1 diabetes in a random-order crossover study under real-world conditions. The study will assess the safety and reliability of both iLet configurations. Our primary objective is to assess whether the iLet operates as designed comparing the insulin-only configuration of the Gen 3.2 iLet bionic pancreas system with the bihormonal configuration of the device using dasiglucagon at a concentration of 4 mg/ml. Our secondary objective is to assess the impact of both configurations of the Gen 3.2 iLet bionic pancreas system on glycemic control, quality of life, and treatment satisfaction among study participants, their caregivers, partners, and/or family members. The study follows a 2-treatment, 2-period crossover design, 2 and will consist of two 7-day study arms in random order: one bihormonal bionic pancreas arm using insulin lispro or insulin aspart and dasiglucagon, and one insulin-only bionic pancreas arm using insulin lispro or insulin aspart.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and have had clinical type 1 diabetes for at least one year
2. Diabetes managed using an insulin pump for ≥ 3 months
3. Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the participant and are not expected to affect any outcome of the study, in the judgement of the principal investigator)
4. Willing to wear one Dexcom CGM sensor, and up to two steel cannula infusion sets (6 mm Contact Detach) and change infusion sets frequently (if the subject is known not to tolerate steel infusion sets then a plastic set may be used)
5. Have used a CGM for at least one cumulative month over the last 24 months
6. Willing to stay within a 250-mile radius of the designated base throughout the study. Air travel is not permitted.
7. Informed consent obtained before any trial-related activities
8. Have a designated contact (an adult ≥ 18 years of age) willing to serve as an emergency contact for them throughout the study.

Exclusion Criteria:

1. Unable to provide informed consent (e.g. impaired cognition or judgment)
2. Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the iLet, impaired memory, unable to speak and read English)
3. Current participation in another clinical trial with administration of investigational drug.
4. Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the participant
5. Previous exposure to dasiglucagon (otherwise known as ZP4207)
6. Pregnant (positive urine HCG), breast feeding, plan to become pregnant in the next 12 months, or sexually active without use of contraception

   1. Subjects must use acceptable contraception for the two weeks prior to the study, throughout the study and for the two weeks following the study.
   2. Acceptable contraception methods include:Oral contraceptive pills (OCP), Intrauterine Device (IUD, hormonal or copper), Male condoms, Female condoms, Diaphragm or cervical cap with spermicide, Contraceptive patch (such as OrthoEvra), Contraceptive implant (such as Implanon, Nexplanon), Vaginal ring (such as Nuvaring), Progestin shot (such as Depo-Provera), Male partner with a vasectomy proven to be effective by semen analysis
7. Current alcohol abuse (intake averaging >4 drinks daily in last 30 days) or other substance abuse (use within the last 3 months of controlled substances other than marijuana without a prescription)
8. Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
9. Renal failure on dialysis
10. History of cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma, or history of complete pancreatectomy
11. Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. exercise of intensity up to 6 METS) despite medical management, or within the last 12 months before screening a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
12. Abnormal EKG consistent with increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, proximal LAD critical stenosis (Wellen's sign), or prolonged QT interval (> 440 ms). Other EKG findings, including stable Q waves, are not grounds for exclusion as long as the participant is not excluded according to other criteria. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
13. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV
14. History of TIA or stroke in the last 12 months
15. History of liver disease that is expected to interfere with the anti-hypoglycemic action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (e.g. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion.
16. Personal history of pheochromocytoma, MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease

    a.Fractionated metanephrines will be tested to rule out pheochromocytoma in patients with symptoms that could be related to a catecholamine secreting tumor, including those with: Episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension, Paroxyms of tachycardia, pallor or headache
17. History of adrenal disease or tumor that has not undergone characterization for endocrine function
18. Hypertension with systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg despite treatment
19. Recent history of diabetic ketoacidosis (DKA) or severe hypoglycemia in the last 6 months. Severe hypoglycemia is defined as an event that required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma.
20. History of more than 1 episode of DKA requiring hospitalization in the last 2 years
21. History of more than 1 episode of severe hypoglycemia in the last year.
22. Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
23. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
24. Unable or unwilling to completely avoid acetaminophen for duration of study
25. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
26. History of adverse reaction to glucagon (including allergy) besides nausea or vomiting
27. History of severe hypersensitivity to milk proteins or lactose
28. History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
29. Current or planned use of SGLT2 inhibitors (prior use more than 3 months prior to enrollment is acceptable; SGLT2 inhibitors should not be initiated during the trial)
30. If using GLP1, pramlintide, or metformin must be on a stable dose for 3 months prior to enrollment (these agents should not be initiated during the trial)
31. Required use of 2 or more steroid bursts in the 6 months prior to the trial
32. History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
33. Any factors that, in the opinion of the site principal investigator or clinical protocol chair, would interfere with the safe completion of the study, including medical conditions that may require hospitalization during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Castellanos LE, Balliro CA, Sherwood JS, Jafri R, Hillard MA, Greaux E, Selagamsetty R, Zheng H, El-Khatib FH, Damiano ER, Russell SJ. Performance of the Insulin-Only iLet Bionic Pancreas and the Bihormonal iLet Using Dasiglucagon in Adults With Type 1 Diabetes in a Home-Use Setting. Diabetes Care. 2021 Jun;44(6):e118-e120. doi: 10.2337/dc20-1086. Epub 2021 Apr 27. No abstract available. PMID 33906916

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 were ineligible due to lacking a designated contact or were taking arrhythmogenic medications
Groups:
- Bihormonal iLet Bionic Pancreas First, Then Insulin-Only: Each sequence of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or dasiglucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM).
  For this sequence, participants first used the bihormonal iLet bionic pancreas for 1 week. They then used the insulin-only iLet bionic pancreas for 1 week without a washout period.
- Insulin-Only iLet Bionic Pancreas First, Then Bihormonal: Each sequence of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or dasiglucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM).
  For this sequence, participants first used the insulin-only iLet bionic pancreas for 1 week. They then used the bihormonal iLet bionic pancreas for 1 week without a washout period.
Period: Overall Study
Arm/Group | Bihormonal iLet Bionic Pancreas First, Then Insulin-Only | Insulin-Only iLet Bionic Pancreas First, Then Bihormonal
Started | 5 | 5
Completed (This is a crossover study. All subjects will participate in both arms.) | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each sequence of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or dasiglucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM).
  Participants were randomized to either first use the bihormonal iLet bionic pancreas for 1 week followed by the insulin-only iLet bionic pancreas for 1 week or to first use the insulin-only iLet bionic pancreas for 1 week followed by the bihormonal iLet for 1 week.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time That Valid CGM Glucose Readings Are Captured by the iLet Bionic Pancreas
Description: Goal for the percentage of time that valid CGM glucose readings are captured by the iLet is ≥80%.
Time Frame: Days 1-7
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Bihormonal iLet Bionic Pancreas: Each arm of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or glucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM). For the purposes of this study, this study arm will use insulin and dasiglucagon in the Bihormonal iLet Bionic Pancreas.
  Bihormonal iLet Bionic Pancreas: Bihormonal iLet Bionic Pancreas using insulin and dasiglucagon
  Dasiglucagon: Experimental stable glucagon for use in the iLet Bionic Pancreas
- Insulin-Only iLet Bionic Pancreas: Each arm of the study will use the iLet Bionic Pancreas. The iLet is an autonomous infusion pump controlled by the bionic pancreas control algorithm that calculates and doses insulin and/or glucagon based on glucose values received by the Dexcom G5 Continuous Glucose Monitor (CGM). For the purposes of this study, this study arm will use just insulin in the Insulin-only iLet Bionic Pancreas.
  Insulin-only Bionic Pancreas: Insulin-only iLet Bionic Pancreas using just insulin
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
percentage of time | 89.2 (6.4) | 91.0 (6.4)

2. Primary Outcome: Percentage of Time That Each Drug Channel of the iLet Bionic Pancreas is Available
Description: Goal for the percentage of the time that each drug channel (insulin, and if applicable, glucagon) is available is ≥95%.
Time Frame: Days 1-7
Population: Percent of time that insulin channel available measured in both groups. Percent of time that glucagon channel available measured only in bihormonal group.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
percentage of time
  % of time that insulin channel available | 99.1 (1.3) | 99.7 (0.20)
  % of time that glucagon channel available: number analyzed (Participants) | 10 | 0
  % of time that glucagon channel available | 99.7 (0.37) |

3. Primary Outcome: The Ratio of Cumulative Drug Doses Delivered to Cumulative Drug Doses Attempted for Insulin and Dasiglucagon
Description: Goal for the ratio of cumulative drug doses delivered to cumulative drug doses attempted is between 0.95 and 1.05, inclusive, for insulin and, if applicable, for glucagon.
Time Frame: Days 1-7
Population: Ratio of cumulative insulin doses delivered to cumulative insulin doses attempted was measured in both groups. Ratio of cumulative glucagon doses delivered to cumulative glucagon doses attempted only measured in bihormonal arm.
Measure: Mean (Standard Deviation); unit: ratio of dose delivered:dose attempted
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
ratio of dose delivered:dose attempted
  Ratio for insulin | 0.999 (0.006) | 1.002 (0.004)
  Ratio for glucagon: number analyzed (Participants) | 10 | 0
  Ratio for glucagon | 1.019 (0.002) |

4. Secondary Outcome: Proportion of Time With CGM Glucose < 54 mg/dl
Time Frame: Days 2-7
Measure: Median (Inter-Quartile Range); unit: proportion of time
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
proportion of time | 0.2 [0 to 0.3] | 0.6 [0.2 to 1.1]

5. Secondary Outcome: Mean Continuous Glucose Monitor Glucose Concentration
Description: Mean continuous glucose monitor glucose concentration measured days 2-7
Time Frame: Days 2-7
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
mg/dl | 139 (11) | 149 (13)

6. Secondary Outcome: Proportion of Time Across Days 2-7 Within the CGM Glucose Range of 70-180 mg/dl
Time Frame: Days 2-7
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
percentage of time | 79 (9) | 71 (8)

7. Secondary Outcome: Mean Grams of Carbohydrate Per Day to Treat or Prevent Hypoglycemic Events (Reported Daily by Subjects)
Time Frame: Days 1-7
Measure: Mean (Standard Deviation); unit: grams of carbs per day
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
Number analyzed (Participants) | 10 | 10
grams of carbs per day | 18 (21) | 16 (13)

ADVERSE EVENTS:
Time Frame: After the 14-day treatment period, two follow-up visits were required; the first in 10 (±3) days and the second in 25 (±4) days after the end of the intervention period (day 14).
Arm/Group | Bihormonal iLet Bionic Pancreas | Insulin-Only iLet Bionic Pancreas
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bihormonal iLet Bionic Pancreas (N=10) | Insulin-Only iLet Bionic Pancreas (N=10)
Nausea (Gastrointestinal disorders) | 4 | 3
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT03840278/Prot_SAP_000.pdf